CLINICAL TRIAL: NCT06949124
Title: A Single-center, Single-arm, Open-label, Fixed-sequence, Self-controlled Clinical Study to Evaluate the Effects of SHR7280 on the Pharmacokinetics of SHR7280 and Midazolam, S-warfarin, Omeprazole, Digoxin, and Rosuvastatin in Healthy Subjects
Brief Title: A Phase 1 Clinical Study to Evaluate the Effects of SHR7280 on the Pharmacokinetics of Midazolam, S-warfarin, Omeprazole, Digoxin, and Rosuvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR7280-108
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis; Uterine Fibroids; Assisted Reproduction
MeSH Terms: conditions — Endometriosis; Leiomyoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: SHR7280 Tablets

INTERVENTIONS:
Drug: SHR7280 Tablets — SHR7280 tablets.

SUMMARY:
The purpose of this study is to evaluate the effects of SHR7280 on the pharmacokinetics of midazolam, S-warfarin, omeprazole, digoxin and rosuvastatin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form prior to any study-related activities, understand the procedures and methods of the study, and agree to complete this study in strict accordance with the clinical study protocol.
2. Males aged 18-45 years (inclusive).
3. Subjects who are generally healthy as judged by the investigator based on medical history, vital signs, physical examination, laboratory tests, and electrocardiogram (ECG).
4. Weight ≥ 50 kg and body mass index (BMI) : 19-26 kg/m2 (inclusive).
5. Informed consent was obtained and patients did not plan to have children within 3 months after the last dose of medication, and they agreed to use highly effective contraception.

Exclusion Criteria:

1. Those with clinically significant abnormalities in physical examination, vital signs (respiration, temperature, pulse), other laboratory tests, chest imaging, abdominal ultrasound, etc.
2. Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody and syphilis antibody positive.
3. Patients with any previous diseases that increase the risk of bleeding.
4. Patients with previous chronic or severe medical history or existing diseases of the respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, and mental system, who were judged by the investigators to be not suitable for the trial.
5. History of blood donation or blood loss ≥ 400 mL or blood transfusion within 3 month before screening.
6. Subjects with other factors considered by the investigator to be ineligible for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | 0 to anticipated 29 days.
Area under the curve from time 0 to infinity (AUC0-∞) | 0 to anticipated 29 days.
Area under the curve from time 0 to time t (AUC0-t) | 0 to anticipated 29 days.

SECONDARY OUTCOMES:
Time to reach the maximum concentration (Tmax) | 0 to anticipated 29 days.
Half-life (t1/2) | 0 to anticipated 29 days.
Apparent clearance (CL/F) | 0 to anticipated 29 days.
Adverse events (AEs) | Baseline up to Day 29.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided